CLINICAL TRIAL: NCT06237738
Title: The Effect of Stress Ball Use on Invasive Pain Associated With Cannulation in Hemodialysis Patients: A Randomized, Controlled, Single-Blind Study
Brief Title: Impact of Stress Balls on Cannulation Pain in Hemodialysis: A Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, BETÜL TOSUN, PhD, Associate Professor, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-64
Record Dates: First submitted 2024-01-12; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Pain; Cannula Site Pain
Keywords: Pain Management; Renal Dialysis; Cannulation; Arteriovenous Fistula; Pain Measurement
MeSH Terms: conditions — Pain; Agnosia; Arteriovenous Fistula

STUDY DESIGN:
Intervention Model Description: This single-blind, randomized, controlled clinical trial evaluated the effectiveness of stress balls in alleviating cannulation-related pain in adults undergoing hemodialysis. The study, which targeted a sample size of 64 based on G*Power analysis for a 95% confidence interval and 80% power with an expected effect size of 0.68, successfully distributed participants into two equal groups of 32: an experimental group and a control group. Participants, aged 18 and above and experiencing a pain level of 1 or more on the Visual Analog Scale (VAS), were randomly assigned to either group. The experimental group utilized stress balls in their non-cannulating hand for three minutes before cannulation during their Monday, Wednesday, and Friday sessions, while the control group, attending on Tuesday, Thursday, and Saturday, received standard care. Data collection encompassed VAS pain level measurements and socio-demographic and medical information gathered via a semi-structured questionnaire.
Who Masked: Investigator
Masking Description: This study employs a single-blind design. In this setup, the participants are unaware of their group allocation, meaning they do not know whether they are in the intervention group (receiving the stress balls) or in the control group (receiving standard care without any additional intervention). The researchers and healthcare professionals administering the treatment are aware of each participant's group assignment. This approach ensures that the participants' responses and reported outcomes, such as pain levels measured by the Visual Analog Scale (VAS), are not influenced by their knowledge of the treatment received. The single-blind design is chosen to maintain the objectivity of the participants' responses while allowing the healthcare team to appropriately administer and monitor the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Ball Intervention (Experimental): Participants in this group were provided with stress balls to use during their hemodialysis sessions, specifically before the cannulation process. These stress balls, made from medium-firm, high-quality silicone, were utilized by squeezing with the hand opposite the one receiving cannulation. This activity, performed three minutes before the cannulation, aimed to reduce the levels of pain experienced by the participants. The use of stress balls was integrated into the regular hemodialysis routine, and participants consistently engaged in this practice before each cannulation over the course of the study. This intervention provided valuable insights into the effectiveness of simple, non-pharmacological methods for pain management in a clinical setting.
  Interventions: Behavioral: Stress Ball Use
- Standard Care Control (No Intervention): Participants in the control group did not receive any additional intervention. They continued to receive standard care during their hemodialysis sessions, without the use of any extra tools like stress balls for pain management. This group served as a comparison point to assess the effectiveness of the intervention implemented in the experimental group. By maintaining their routine hemodialysis care, the control group provided essential data for evaluating the impact of the stress ball intervention. The completion of their participation in the study was crucial in establishing a baseline for pain levels during cannulation without any non-pharmacological interventions.

INTERVENTIONS:
Behavioral: Stress Ball Use — The intervention in this study involves the use of stress balls provided to participants in the intervention group. These are specially designed medium-firm silicone balls intended for squeezing with the hand opposite the one receiving cannulation during hemodialysis sessions. The primary objective of this intervention is to offer a simple, non-pharmacological method to potentially alleviate the pain associated with the cannulation process. Participants are instructed to use the stress ball for a period of three minutes before the start of cannulation. This activity is hypothesized to focus the participant's attention and possibly reduce the perception of pain, contributing to a more comfortable and less distressing cannulation experience.
  Arms: Stress Ball Intervention

SUMMARY:
Background: Chronic kidney disease significantly impacts patients and their families, with a portion requiring hemodialysis. Hemodialysis involves repeated vascular cannulation, often causing moderate to severe pain. This planned study aims to investigate the efficacy of using stress balls as a non-pharmacological intervention to reduce pain during cannulation in hemodialysis patients.

Methods: This upcoming single-blind, randomized, controlled trial will involve 64 adult patients undergoing hemodialysis, divided equally into an intervention group and a control group. The intervention group will use stress balls during cannulation, while the control group will receive standard care. Pain levels will be assessed using the Visual Analog Scale (VAS), and additional socio-demographic and medical data will be collected through a semi-structured questionnaire.

Objectives: The primary objective of this proposed study is to evaluate the effectiveness of stress balls in reducing pain associated with cannulation in hemodialysis patients. The study also aims to contribute to pain management strategies in this patient population.

Ethical Considerations: The study will adhere to the Helsinki Declaration principles and will seek approval from the local ethics committee. Informed consent will be obtained from all participants, and the study's design, methodology, and ethical standards will be transparently registered on ClinicalTrials.gov prior to commencement.

Statistical Analysis: Data analysis will be planned using JAMOVI software. The primary analysis will compare VAS scores between groups and over time using Robust ANOVA, with adjustments for multiple comparisons.

Significance: This planned study addresses the need for non-pharmacological pain management during hemodialysis cannulation. The findings are expected to enhance patient comfort and adherence to dialysis regimens, ultimately improving their quality of life.

Background: Chronic kidney disease (CKD) has a significant impact on patients and their families, with many eventually requiring hemodialysis treatment. Hemodialysis often involves repeated vascular cannulation, which can cause moderate to severe pain. This study has been conducted to investigate the efficacy of using stress balls as a non-pharmacological intervention to reduce pain during cannulation in hemodialysis patients.

Methods: In this completed single-blind, randomized, controlled trial, 64 adult patients undergoing hemodialysis were divided into two groups. The intervention group used stress balls during cannulation, while the control group received standard care without the use of stress balls. Pain levels were assessed using the Visual Analog Scale (VAS). Additionally, socio-demographic and medical data were collected through a semi-structured questionnaire.

Objectives: The primary objective of the study was to evaluate the effectiveness of stress balls in reducing pain associated with cannulation in hemodialysis patients. The study also aimed to contribute to the development of pain management strategies for this patient population.

Ethical Considerations: The study adhered to the principles of the Helsinki Declaration and received approval from the local ethics committee. Informed consent was obtained from all participants, ensuring transparency about the study's purpose, processes, and potential risks.

Statistical Analysis: Data from the study were analyzed using JAMOVI software. The primary analysis involved comparing VAS scores between the intervention and control groups over time using Robust ANOVA, with adjustments for multiple comparisons.

Significance: The study addressed the need for non-pharmacological pain management methods during hemodialysis cannulation.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a critical health issue globally, affecting millions. Many CKD patients require hemodialysis, involving arteriovenous fistula cannulation, which often leads to moderate to severe pain. This pain can negatively impact patient compliance and quality of life. Recognizing the potential benefits of non-pharmacological interventions, this study was conducted to evaluate the effectiveness of stress balls in reducing pain experienced during cannulation in hemodialysis patients.

The primary objective of this completed study was to determine whether the use of stress balls during cannulation significantly reduces pain levels in hemodialysis patients, as measured by the Visual Analog Scale (VAS).

In this single-blind, randomized, controlled trial conducted at a state hospital's hemodialysis unit in Turkey, 64 adult patients undergoing hemodialysis were enrolled. These patients, all with a VAS score of 1 or higher, were randomly assigned to either an intervention group (using stress balls during cannulation) or a control group (receiving standard care). The intervention group included patients attending sessions on Monday, Wednesday, and Friday, while the control group comprised those attending on Tuesday, Thursday, and Saturday. The intervention involved using the stress ball in the non-cannulated hand for three minutes before cannulation.

Pain levels were measured using the VAS at each of the 12 sessions of cannulation for every patient, providing comprehensive data on pain levels. A semi-structured questionnaire was used to collect socio-demographic and medical data. The data were analyzed using JAMOVI software, with Robust ANOVA employed for comparisons.

The study adhered strictly to the Helsinki Declaration's principles. Ethical approval was obtained from the local ethics committee, and informed consent was secured from all participants. The study's design, methodology, and ethical considerations were transparently registered on ClinicalTrials.gov.

The study hypothesized that the use of stress balls would lead to a significant reduction in pain levels during cannulation. This intervention was expected to provide a simple, cost-effective, and accessible method to enhance patient comfort and adherence to hemodialysis, thereby improving their overall quality of life.

The results of this study could significantly contribute to improved pain management strategies for hemodialysis patients. Demonstrating the efficacy of stress balls as a non-pharmacological intervention could offer a straightforward, economical, and accessible approach to enhancing patient comfort during hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older)
* Visual Analog Scale (VAS) score of 1 or higher
* Willingness to participate in the study

Exclusion Criteria:

* Individuals with communication barriers such as severe hearing or cognitive impairments
* Patients with issues in the arm/hand where the stress ball would be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Pain Level Reduction Title: Pain Level Reduction Pain Level Reduction | Hemodialysis patients were monitored over a period of one month, encompassing twelve sessions.
  The primary outcome measure was the reduction in pain levels as assessed by the Visual Analog Scale (VAS). This measure evaluated the effectiveness of the stress ball intervention in reducing the pain experienced by participants during the cannulation process in hemodialysis sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- 25 Aralik State Hospital, Gaziantep, Sahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tosun B, Berse S, Dirgar E, Ozen N. Effect of stress ball use on cannulation-related invasive pain in Hemodialysis patients: a randomized controlled, single-blind study. BMC Nephrol. 2025 Mar 20;26(1):140. doi: 10.1186/s12882-025-04071-w. PMID 40114094